CLINICAL TRIAL: NCT07284472
Title: Phase 2/3, Double-blind, Placebo-controlled Study to Evaluate the Safety and Efficacy of EXV-802 and EXV-801 in the Treatment of Agitation in Participants With Alzheimer's Disease Dementia
Brief Title: Safety and Efficacy of EXV-802 and EXV-801 in the Treatment of Agitation in Alzheimer's Disease Dementia
Acronym: SERENADA
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Exciva GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EXV802-2-1; 2024-517388-22-00 (EU CTIS Number)
Record Dates: First submitted 2025-11-27; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Agitation Associated With Alzheimer's Disease Dementia
MeSH Terms: interventions — Dextromethorphan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- EXV-802 (Experimental)
  Interventions: Drug: EXV-802
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- EXV-801 (Experimental)
  Interventions: Drug: EXV-801

INTERVENTIONS:
Drug: EXV-802 — Specified dose twice daily
  Other Names: Dextromethorphan + EXV-801
  Arms: EXV-802
Drug: Placebo — Specified dose twice daily
  Arms: Placebo
Drug: EXV-801 — Specified dose twice daily
  Arms: EXV-801

SUMMARY:
The goal of this clinical trial is to learn if the investigational drugs EXV-802 and EXV-801 can safely and effectively reduce agitation in participants with Alzheimer's Disease Dementia.

Researchers will compare EXV-802 and EXV-801 with a placebo to see if EXV-802 and/or EXV-801 reduces agitation more effectively than the placebo.

ELIGIBILITY:
Inclusion criteria:

1. The participant is an adult male or female between the ages of 55 to 90 years inclusively, who can move around by themselves, with a walker, or with a wheelchair.
2. A previously established diagnosis of AD dementia.
3. The participant meets definition for agitation which require treatment with medicines.
4. The severity of agitation is at least moderate.

Exclusion criteria:

1. The participant has a confirmed primary diagnosis of a dementia-related disease other than AD dementia.
2. The participant has symptoms of agitation that are due to psychiatric conditions other than AD dementia.
3. The participant has a history of uncontrolled seizures or a history of epilepsy.
4. The participant lacks a caregiver or support person who attends regularly to the participants' needs.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline to endpoint (Week 6) in the Cohen-Mansfield Agitation Inventory (CMAI) score (range 1 - 7 per item; higher scores indicate more severe agitation) | At Week 6

SECONDARY OUTCOMES:
Changes from baseline to endpoint (Week 6) in the Clinical Global Impression - Severity (CGI-S) scale score (range 1 - 7; higher scores indicate worse disease severity) | At Week 6

OTHER OUTCOMES:
Changes from baseline to endpoint (Week 6) in the Neuropsychiatric Inventory - Clinician Rating (NPI-C) Caregiver Distress score for agitation and aggression (range 0 - 5 per item; higher scores indicate greater caregiver distress) | At Week 6
Changes from baseline to endpoint (Week 6) in the Neuropsychiatric Inventory - Clinician Rating (NPI-C) Irritability/Liability score (range 0 - 12 per item composite; higher scores indicate greater symptom severity) | At Week 6
Changes from baseline to endpoint (Week 6) in the Neuropsychiatric Inventory - Clinician Rating (NPI-C) Sleep Disorders score (range 0 - 12 per item composite; higher scores indicate worse sleep disturbance) | At Week 6

IPD SHARING:
Plan to Share IPD: Undecided